CLINICAL TRIAL: NCT02221986
Title: Interdisciplinary Rehabilitation of Patients With Glioma During Anti-cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Anders Hansen, Physiotherapist, Master of Health Science, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20140108
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2017-09

CONDITIONS: Neoplasms; CNS Neoplasms
Keywords: Interdisciplinary rehabilitation; Neurooncology; Physiotherapy; Occupational therapy; Neurorehabilitation; Glioma
MeSH Terms: conditions — Neoplasms; Central Nervous System Neoplasms; Glioma

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Interdisciplinary rehabilitation (Experimental): The intervention consists of 6 weeks intensive outpatient physiotherapy in conjunction with 0-6 weeks of occupational therapy if need is indicated. The physical intervention contains supervised group exercise of 90 minutes three times a week in groups up to four patients included continuously.
  The occupational therapy intervention consists of individual training 60 minutes twice a week for patients having deficits in activity or participation levels measured by the Assessment of Motor and Process Skills (AMPS).
  Interventions: Behavioral: Interdisciplinary rehabilitation
- Care as usual (No Intervention): The control group receives usual standard of care (e.g. no training, individual training or group training in the municipality). The amount of training in this group is based on a questionnaire at the follow-up trials.

INTERVENTIONS:
Behavioral: Interdisciplinary rehabilitation
  Arms: Interdisciplinary rehabilitation

SUMMARY:
The results of the present RCT study will add to the growing body of literature investigating the potential role of exercise as a supportive therapeutic intervention for patient with glioma.

DETAILED DESCRIPTION:
Gliomas are the most frequent primary neoplasm in the CNS and according to the World Health Organization histologically categorized into low-grade glioma (LGG) (WHO grades I/II) or high-grade glioma (HGG) (WHO grades III/IV). Gliomas are among the biggest challenges within the field of neuro-rehabilitation and oncology, and optimising treatment by improving QoL, function and cognition is of major clinical importance in this population. Because the majority of patients cannot be cured, clinical cancer research traditionally have focused on prolonging survival, exposing relapse or optimising the response to the medical treatment. Today there is a general consensus that health-related quality of life (HRQoL) is important in the evaluation of new treatments. However, research in HRQoL among patients with gliomas is scarce compared to the other categories of patients with tumors. In recent years have exercise become an important part of cancer treatment. The effects is well documented in studies among other cancer patients than gliomas and includes improvements of quality of life, physical function, reduce fatigue and thereby supports daily activities among cancer patients'. Inpatient rehabilitation studies among glioma patients have also indicated improved HRQoL and functional measurements such as activity of daily life, mobility and cognition. Despite of this rehabilitation efforts is still not emphasized in this population and recent literature concludes that there are no well-designed clinical studies examining the effect of multidisciplinary rehabilitation among Glioma patients. This study is the first to investigate the effect of an intensive specialised interdisciplinary outpatient rehabilitation program among gliomas patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary glioma (WHO grades I-IV)
* Age ≥ 18
* Reference with diagnosis or treatment at Odense University Hospital
* Karnofsky performance score (KPS) ≥70
* Ability to understand Danish.

Exclusion Criteria:

* Pregnancy
* Known psychiatric diagnosis or substance abuse
* Heart problems excluding intense exercise (NYHA group III and IV)
* Pronounced impressive/expressive aphasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | Change from Baseline HRQoL at 6 months
  Questionnaires EORTC-QLQ-30 & BN-20

SECONDARY OUTCOMES:
Symptom burden | Change from Baseline Symptom burden at 6 months
  Assessed through EORTC-QLQ-30 & BN-20
Physical activity levels | Change from Baseline Physical activity levels at 6 months
  Physical activity at work and leisure time ( Assessed through questionnaire by Saltin and Grimsby 1968 and Physical Activity Scale)
Muscle strength | Change from Baseline Musclestrength at 3 months
  Assessed through 3-8 submax repetition maximum
VO2peak | Change from Baseline VO2peak at 3 months
  Assessed through Åstrand 1-pkt. cycle test.
Balance | Change from Baseline Balance at 3 months
  Assessed through wii balance board
Gait function | Change from Baseline gait function at 3 months
  Assessed through 10 meter walk test. Time and step frequency.
Activity levels | Change from Baseline Activity levels at 3 months
  Assessed through questionnaire (Impact on Participation and Autonomy)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Søgaard, Professor, Study Chair — University of Southern Denmark
Locations (1):
- Odense University Hospital, Odense, Funen, Denmark

REFERENCES:
- [Derived] Hansen A, Pedersen CB, Jarden JO, Beier D, Minet LR, Sogaard K. Effectiveness of Physical Therapy- and Occupational Therapy-Based Rehabilitation in People Who Have Glioma and Are Undergoing Active Anticancer Treatment: Single-Blind, Randomized Controlled Trial. Phys Ther. 2020 Mar 10;100(3):564-574. doi: 10.1093/ptj/pzz180. PMID 32043148
- [Derived] Fahrenholtz ML, Hansen A, Sogaard K, Andersen LN. Finding 'the inner drive' for a rehabilitation process: a small-scale qualitative investigation among male patients with primary glioma. BMJ Open. 2019 Dec 8;9(12):e031665. doi: 10.1136/bmjopen-2019-031665. PMID 31818840
- [Derived] Hansen A, Rosenbek Minet LK, Sogaard K, Jarden JO. The effect of an interdisciplinary rehabilitation intervention comparing HRQoL, symptom burden and physical function among patients with primary glioma: an RCT study protocol. BMJ Open. 2014 Oct 3;4(10):e005490. doi: 10.1136/bmjopen-2014-005490. PMID 25280804